CLINICAL TRIAL: NCT04994002
Title: A Phase 1b, Open-Label, Pharmacokinetic, Pharmacodynamic, Safety and Tolerability Study of CERC-006 in Adults (Aged 18-31 Years) With Complex Lymphatic Malformations
Brief Title: A Pharmacokinetic, Pharmacodynamic, Safety and Tolerability Study of CERC-006 in Adults With Complex Lymphatic Malformations
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CERC-006-LM-101
Record Dates: First submitted 2021-07-20; First posted 2021-08-06 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Lymphatic Malformation
Keywords: Lymphatic Malformation; Complex Lymphatic Malformations; CERC-006
MeSH Terms: conditions — Lymphatic Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: CERC-006 (0.5 mg) (Experimental): Approximately 5 participants will receive CERC-006 at a dose of 0.5 mg twice daily for 28 days.
  Interventions: Drug: CERC-006
- Cohort 2: CERC-006 (1 mg) (Experimental): Following a safety review, if there are no clinically important safety findings in Cohort 1, a second cohort of approximately 5 participants will be enrolled to receive CERC-006 at a dose of 1 mg twice daily for 28 days.
  Interventions: Drug: CERC-006

INTERVENTIONS:
Drug: CERC-006 — Oral solution

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of CERC-006 in adults (aged 18-31 years) with active, moderate to severe complex lymphatic malformations.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill the following requirements to be eligible for the study:

1. Participant is 18 to 31 years of age (inclusive) at the time of consent.
2. Participant has a verified diagnosis of a complex lymphatic malformation. Other moderate to severe vascular anomalies with associated lymphatic involvement will be considered, with approval by the study medical monitor.
3. Participant's complex lymphatic malformation is considered, in the opinion of the investigator, to be moderate to severe.
4. Participant has adequate liver function defined as:

   * Total bilirubin (sum of conjugated and unconjugated) ≤1.5 × upper limit of normal (ULN)
   * Aspartate transaminase/Alanine aminotransferase (AST/ALT) <5 × ULN
   * Serum albumin > 2 g/dL
5. Participant has fasting low-density lipoprotein (LDL) of <160 mg/dL.
6. Participant has adequate bone marrow function defined as:

   * Peripheral absolute neutrophil count (ANC) > 1000/µL
   * Hemoglobin > 8.0 g/dL
   * Platelet count ≥ 50,000/µL
7. Participant has adequate renal function defined as:

   • Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance of > 50 mL/min according to the Cockcroft-Gault equation
8. Participant has agreed to and met the washout period as follows:

   * At least 14 days prior to initiation of CERC-006 if receiving sirolimus (also known as rapamycin), mitogen-activated protein kinase (MEK) inhibitors, phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) inhibitors, interferon alfa 2b, vascular endothelial growth factor receptor 3 (VEGFR-3) inhibitors, and/or other systemic agents targeting lymphatic malformation
   * At least 7 days prior to initiation of CERC-006 if receiving topical agents targeting lymphatic malformation
9. Participant has a Karnofsky performance status of ≥50%.

Exclusion Criteria:

The presence of any of the following criteria excludes a participant from the study:

1. Participant has a concurrent severe or uncontrolled medical disorder, which could compromise participation in the study.
2. Participant has significant impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of CERC-006.
3. Participant has taken any medication that is a strong cytochrome P450 3A4 (CYP3A4) enzyme inducer or inhibitor within 2 weeks prior to first dose of study drug, or in the opinion of the Investigator, subject may require such medication during the study
4. Participant is receiving chronic treatment with systemic steroids or another immunosuppressive agent, or in the opinion of the Investigator, subject may require such medication during the study
5. Participant has undergone myelosuppressive chemotherapy within 2 weeks, or radiation within 4 weeks prior to first dose of study drug.
6. Participant has a known history of uncontrolled hypertension, cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, cardiac conduction problems, heart failure, exercise-related cardiac events including syncope and pre-syncope, or a known family history of sudden cardiac death or ventricular arrhythmia.
7. Participant has received treatment with a medication that has the potential to prolong the QT interval within 1 week prior to the first dose of study drug, or in the opinion of the Investigator, subject may require such medication during the study.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of CERC-006 in Adults (Aged 18-31 Years) with Active, Moderate to Severe Complex Lymphatic Malformations | Up to approximately 6 weeks
  Safety and tolerability will be assessed by incidence of adverse events (AEs). Clinically significant changes from baseline in vital signs, ocular exams, cardiology tests including echocardiogram (ECHO) and electrocardiogram (ECG), and clinical laboratory results will be recorded as AEs.

SECONDARY OUTCOMES:
Serum Concentrations of CERC-006 | Baseline (Day 1) up to 3 days after last dose of study drug (up to approximately 4 weeks)
Change from Baseline in Levels of mTOR Related Pathway Biomarkers | Baseline (Day 1) up to 3 days after last dose of study drug (up to approximately 4 weeks)
Change from baseline to end of treatment in radiologic assessment, if clinically indicated and/or clinical signs/symptoms of disease | Baseline (Screening) up to 3 days after last dose of study drug (up to approximately 8 weeks)
  Radiologic disease assessment will be done if clinically indicated, at the discretion of the investigator.
Change from Baseline in 36-Item Short Form Health Survey (SF-36) Score | Baseline (Day 1) up to 3 days after last dose of study drug (up to approximately 4 weeks)
  SF-36 score will measure eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores on each scale will be directly transformed into a 0-100 scale, where a lower score indicates more disability.
Change from Baseline in Karnofsky Performance Status Score | Baseline (Day 1) up to 3 days after last dose of study drug (up to approximately 4 weeks)
  Karnofsky Performance Status score will be measured on a scale from 0 percent (%) to 100%, where a lower percentage score indicates a worse disease state.
Change from Baseline in Pain Scale Assessment | Baseline (Day 1) up to 3 days after last dose of study drug (up to approximately 4 weeks)
  Pain scale assessment will be done using a 100 mm Visual Analog Scale (VAS) from no pain (0 mm) to extreme pain (100 mm).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No